CLINICAL TRIAL: NCT05360953
Title: Treating Nightmares in Posttraumatic Stress Disorder With the α-adrenergic Agents Clonidine and Doxazosin: A Randomized-Controlled Feasibility Study (ClonDoTrial)
Brief Title: Treating Nightmares in Posttraumatic Stress Disorder With Clonidine and Doxazosin
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to recruitment issues
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Stefan Roepke, Prof. Dr. Stefan Roepke, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ClonDO
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Nightmares; Posttraumatic Stress Disorder; Clonidine; Doxazosin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Clonidine; Doxazosin

STUDY DESIGN:
Intervention Model Description: Randomized controlled study (double-blind)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm Clonidine (Experimental)
  Interventions: Drug: Clonidine
- Arm Doxazosin (Experimental)
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — All patients enrolled establish their individually tolerable dose by dose Titration. Dosage up to a maximum of 0.375 clonidine. Using capsules of 0,075 mg clonidine.
  Arms: Arm Clonidine
Drug: Doxazosin — All patients enrolled establish their individually tolerable dose by dose. Dosage up to a maximum of 10 mg doxazosin. Using capsules of 2 mg doxazosin.
  Titration.
  Arms: Arm Doxazosin
Drug: Placebo — All patients enrolled establish their individually tolerable dose by dose Titration. Dosage up to a maximum of 5 capsules. Using capsules of placebo.
  Arms: Placebo

SUMMARY:
This randomized controlled trial will test the hypothesis that oral Clonidine or Doxazosin improves nightmares (primary outcome), other PTSD symptoms and psychopathology (secondary outcomes) to a greater extent than placebo over a ten week intervention phase in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of posttraumatic stress disorder (PTSD) according to DSM 5 with a 20 item CAPS-5 total score ≥ 26
2. At least two nightmares a week, an intensity score ≥ 2, with a CAPS-IV B2 (frequency and intensity for the last week) score ≥ 5
3. Men and women between 18 and 65 years of age
4. Written informed consent
5. The patient has the capacity to give consent (He/she is able to understand the nature and anticipated effects/side effects of the proposed medical intervention)
6. The patient is not breastfeeding
7. Women of child-bearing potential must have a negative urine or serum pregnancy test
8. All participants must use highly effective contraception
9. The patient received stable pharmacological medication for at least 4 weeks or at least five times the value of a elimination half-life prior to study baseline (any changes in medication dose or frequency of therapy must be answered with no).

Exclusion Criteria:

1. Disturbances of cardiac impulse formation and conduction, for example sick sinus syndrome or atrioventricular block second and third degree
2. Bradycardia, with a heart rate less than 50 beats per minute
3. Current major depressive episode and a MADRS score > 34
4. The patient does have a known allergy, hypersensitivity or contraindication against clonidine, doxazosin, or other types of quinazolines
5. History of severe orthostatic hypotension
6. Benign prostatic hyperplasia and concomitant congestion of the upper urinary tract, chronic urinary tract infection or bladder stones, hypotension (for benign prostate hyperplasia only)
7. Either overflow bladder or anuria with or without progressive renal insufficiency
8. Planned cataract surgery (risk of 'Intraoperative Floppy Iris Syndrome')
9. Intake of phosphodiesterase-5-inhibitors
10. Intake of methylphenidate
11. Severe hepatic impairment (ASAT or ALAT greater than two times normal)
12. Acute or unstable medical illness
13. Known HIV- and/or active Hepatitis-B- or Hepatitis-C-infection
14. Current or past malignant illness
15. The patient does have clinically significant abnormalities in 12-lead ECG
16. The patient does have clinically significant laboratory abnormalities
17. Epilepsy
18. Dementia
19. Current substance/alcohol use disorder (≤ 3 months)
20. Psychotic disorder
21. Bipolar disorder
22. Current anorexia nervosa
23. Acute suicidality (any suicidal ideation of type of 5 in the C-SSRS in the past month)
24. Intake of alpha adrenergic agents (Clonidine, doxazosin, or others) within 4 weeks prior to baseline (randomization)
25. Trauma-focused psychotherapy four weeks before the trial
26. Initiation of sleep medication 4 weeks prior to baseline
27. The patient is unwilling to consent to saving, processing and propagation of pseudonymized medical data for study reasons
28. Patients, who may be dependent on the sponsor, the investigator or the trial sites
29. The patient is legally detained in an official institution
30. The patient did participated in other interventional trials during the 3 months before and at the time of this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of frequency and intensity of nightmares | 10 weeks
  Change of Frequency and intensity of nightmares, measured with the Clinician-Administered PTSD Scale-IV (CAPS-IV) B2 score for the last week, range 0-8, from baseline until directly after last intervention. A lower score indicates less frequent and/or intense nightmares.

SECONDARY OUTCOMES:
Change of frequency and intensity of nightmares | 1,2,3,4,5,6 and 8 weeks
  Change of Frequency and intensity of nightmares, measured with the Clinician-Administered PTSD Scale-IV (CAPS-IV) B2 score for the last week, range 0-8, from baseline until directly after last intervention. A lower score indicates less frequent and/or intense nightmares.
Change from baseline of the CLINICIAN-ADMINISTERED PTSD SCALE FOR DSM-5 (CAPS-5) total score | 6 and 10 weeks
  Change from baseline of the CAPS-5 total score (overall PTSD symptoms, last week) (minimum value = 0; maximum value = 80; higher scores indicate higher PTSD symptom severity)
Change from baseline of the Pittsburgh Sleep Quality Index-Addendum for PTSD | 6 and 10 weeks
  Change from baseline of the Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI A) (PTSD related sleep symptoms); (score = 0-21 point, 0 = no difficulty; 21 = severe difficulty in all areas)
Change from baseline of the -Montgomery Asberg Depression Rating Scale (MDRS) | 6 and 10 weeks
  Change from baseline of the MADRS (scores: 0 - 60; 0 - 6 = no depression; 7 - 19 = light depression; 20 - 34 = moderate depression; > 34 severe depression)
Weekly mean of change from baseline of daily total sleep time | during 10 weeks
  Weekly mean of change from baseline of the patients daily total sleep time (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients sleep onset latency at night (in minutes), assessed with sleep diaries | during 10 weeks
  Weekly mean of change from baseline of the patients sleep onset latency at night (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients recuperation of night sleep | during 10 weeks
  Weekly mean of change from baseline of the patients recuperation of night sleep (5-point Likert scale, 1 = very much; 5
  = not at all), assessed with sleep diaries
Weekly mean of change from baseline of the patients time awake at night | during 10 weeks
  Weekly mean of change from baseline of the patients time awake at night (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients number of nightmares last night | during 10 weeks
  Weekly mean of change from baseline of the patients number of nightmares last night (0, 1, 3, 4 or more) assessed with sleep diaries
Weekly mean of change from baseline of the patients intensity of nightmares | during 10 weeks
  Weekly mean of change from baseline of the patients intensity of nightmares (5-point Likert scale, 0 = not at all; 5 = extreme) assessed with sleep diaries
Change from baseline of PTSD symptoms assessed with the PTSD Checklist for DSM-5 | 6 and 10 weeks
  Change from baseline of PCL-5 PTSD Checklist for DSM-5; Score can range from 0-80 (higher scores indicate a higher PTSD symptom severity) Score (0 - 80; higher scores indicating higher chance of a possible PTSD diagnosis)
Change from baseline of the Borderline Symptom List 23 (BSL-23) | 6 and 10 weeks
  Change from baseline of the BSL-23 score (Scores can range from 0 to 92; higher scores indicate higher Borderline symptom severity) Scores: 0 - 4 (0 = no Borderline Symptoms; 4 = severe borderline symptoms)
Change from baseline of the Health-Related Quality of Life (EQ-5D) | 6 and 10 weeks
  Change from baseline of the EQ-5D score (score can range from 0-100; with higher scores indicating a better Health Related Quality of Life) Scores = 1-5 (1 = no problems; 5 = extreme problems)
Overall patients status measured by the Patient Global Impression of Change (PGIC) | 6 and 10 weeks
  Overall patients status measured by the PGIC (Scores can range from 0 - 7; with higher scores indicating higher improvement) score: 0 - 7 (0 = disease deterioration; 7 = disease improvement)
Change from baseline of the Social and Occupational Functioning Assessment Scale | 6 and 10 weeks
  Change from baseline of the Social and Occupational Functioning Assessment Scale (SOFAS); Scores can range from 1 - 100, with higher scores indicating better social and occupational functioning
Change from baseline of the Pittsburgh Sleep Quality Index (PSQI) | 6 and 10 weeks
  Change from baseline of the PSQI; Scores can range from 0 to 21, with higher scores indicating lower sleep quality Scores : 0 - 21, lower scores denote a healthier sleep quality
Change from baseline of symptoms of PTSD and complex PTSD according to ICD-11 assessed with the International Trauma Questionnaire (ITQ) | 6 and 10 weeks
  Change from baseline of symptoms of ITQ, dimensional scores can range from 0 - 24, with higher scores indicating highter PTSD symptom severity
  Categorical Scoring:
  For PTSD items, endorsement of a symptom or functional impairment item is defined as a score of 2 or greater.
  The diagnosis of PTSD is indicated based on the following criteria:
  * Question 1 or 2 = one or more items endorsed (re-experiencing)
  * Question 3 or 4 = one or more items endorsed (avoidance)
  * Question 5 or 6 = one or more items endorsed (sense of current threat)
  * Question 7, 8 or 9 = one or more items endorsed (PTSD functional impairment)
Responder analysis: proportion of patients showing improvement in nightmares | 10 weeks
  Responder analysis: proportion of patients showing improvement in nightmares (change from baseline) defined as decrease of CLINICIAN-ADMINISTERED PTSD SCALE FOR DSM-IV (CAPS-IV B2) ≥50% assessed at the end of treatment
  Score: 0 - 8 (higher scores indicate higher frequency and severity of nightmares)
Remitter analysis: proportion of patients showing full remission of nightmares | 10 weeks
  Remitter analysis: proportion of patients showing full remission of nightmares defined as CLINICIAN-ADMINISTERED PTSD SCALE FOR DSM-IV (CAPS-IV B2) = 0, assessed at the end of treatment; 0 = no nightmares (score 0 - 8; higher scores indicate higher frequency and severity of nightmares))

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (5):
- Germany (5):
  - Universitätsklinikum Tübingen, Tübingen, Germany
  - Berlin St. Hedwig, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Klinik für Psychiatrie und Psychotherapie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim

REFERENCES:
- [Derived] Roepke S, Schoofs N, Priebe K, Wuelfing F, Roehle R, Maslahati T, Stieglbauer K, Biedermann S, Schaefer I, Gallinat J, Ethofer T, Fallgatter AJ, Hanewald B, Mulert C, Schmahl C, Otte C, Koglin S. Treating nightmares in post-traumatic stress disorder with the alpha-adrenergic agents clonidine and doxazosin: protocol for a phase II randomised, double-blind, placebo-controlled parallel-group study (ClonDoTrial). BMJ Open. 2025 Aug 5;15(8):e098161. doi: 10.1136/bmjopen-2024-098161. PMID 40764082